CLINICAL TRIAL: NCT05419804
Title: Placenta Accreta; Total Lower Uterine Segmentectomy With Cervico-corporeal Anastomosis, a Feasibility Study
Brief Title: Placenta Accreta; Total Lower Uterine Segmentectomy With Cervico-corporeal Anastomosis
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Naglaa Mohamed, Principal investigator, Assiut University
Other Study IDs: TLUSCCA
Record Dates: First submitted 2022-05-30; First posted 2022-06-15 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To study feasibility and safety of Total lower uterine segmentectomy with cervico-corporeal anastomosis in conservative management of placenta accreta

DETAILED DESCRIPTION:
Placenta accreta represents a real challenge in modern obstetric care as its incidence is increasing in a parallelism with increased CSs rates. Its management represents another challenge and a multidisciplinary team with clear plans and alternative strategies that fulfill different situation and address different patient needs must be clearly settled in every referral center dealing with placenta accreta.

Hysterectomy without trials of placental separation seems to be the standard and logical procedure. However hysterectomy needs to be a total or at least including the entire invaded Lower uterine segment. Hysterectomy is associated with significant blood loss, and loss of future fertility. There are several fertility conservation approaches with variable success rates, complications, technical demands and costs.

Uterine plication sutures has been reported as successful uterine conservation strategy but subsequent intrauterine adhesions, weak uterine scar and uterine necrosis might culminate in a functionless uterus.

The present work describes total lower uterine segmentectomy with cervical-corporeal anastomosis as a relatively less invasive uterine conservation strategy with minimization of blood loss and transfusion needs. Furthermore, total lower uterine segmentectomy with cervico-corporeal anastomosis has the merits of leaving behind a strong scar and a well-functioning uterus.

ELIGIBILITY:
Inclusion Criteria:

pregnant women diagnosed with placenta accreta by us and Doppler Accreta invading the entire or most of the lus Women who welling uterine conservation, Planned and elective cs for women diagnosed with accreta, and accepting participation

Exclusion Criteria:

women who don't accept participation, women who desire hysterectomy. Women who diagnosed with accrete and placenta separated easily women with concomitant pathology and requiring hysterectomy .

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: pregnant women diagnosed with placenta accreta by us and Doppler Accreta invading the entire or most of the lus Women who welling uterine conservation, planned and elective cs for women diagnosed with accreta, and accepting participation
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Success of procedure | 1year
  Success of procedure regarding ability to preserve the uterus and stoppage of bleeding.
  The bleeding will be evaluated by haemoglobin level preoperative and postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Ezzat H Sayed, professor, Study Chair — Assiut medical school
Locations (1):
- Assiut Medical School, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bloomfield V, Rogers S, Leyland N. Placenta accreta spectrum. CMAJ. 2020 Aug 24;192(34):E980. doi: 10.1503/cmaj.200304. No abstract available. PMID 32839166
- [Background] Zuckerwise LC, Craig AM, Newton JM, Zhao S, Bennett KA, Crispens MA. Outcomes following a clinical algorithm allowing for delayed hysterectomy in the management of severe placenta accreta spectrum. Am J Obstet Gynecol. 2020 Feb;222(2):179.e1-179.e9. doi: 10.1016/j.ajog.2019.08.035. Epub 2019 Aug 27. PMID 31469990
- [Background] Pinas Carrillo A, Chandraharan E. Placenta accreta spectrum: Risk factors, diagnosis and management with special reference to the Triple P procedure. Womens Health (Lond). 2019 Jan-Dec;15:1745506519878081. doi: 10.1177/1745506519878081. PMID 31578123
- [Background] Wortman AC, Alexander JM. Placenta accreta, increta, and percreta. Obstet Gynecol Clin North Am. 2013 Mar;40(1):137-54. doi: 10.1016/j.ogc.2012.12.002. PMID 23466142
- [Background] Society of Gynecologic Oncology; American College of Obstetricians and Gynecologists and the Society for Maternal-Fetal Medicine; Cahill AG, Beigi R, Heine RP, Silver RM, Wax JR. Placenta Accreta Spectrum. Am J Obstet Gynecol. 2018 Dec;219(6):B2-B16. doi: 10.1016/j.ajog.2018.09.042. PMID 30471891
- [Background] Fonseca A, Ayres de Campos D. Maternal morbidity and mortality due to placenta accreta spectrum disorders. Best Pract Res Clin Obstet Gynaecol. 2021 Apr;72:84-91. doi: 10.1016/j.bpobgyn.2020.07.011. Epub 2020 Jul 20. PMID 32778495
- [Background] Biyik I, Keskin F, Keskin EU. Conservative Surgical Treatment of a Case of Placenta Accreta. Rev Bras Ginecol Obstet. 2018 Aug;40(8):494-496. doi: 10.1055/s-0038-1668528. Epub 2018 Aug 24. PMID 30142668
- [Background] Haunschild C, Yeaton-Massey A, Lyell DJ. Antenatal Management of Placenta Accreta. Clin Obstet Gynecol. 2018 Dec;61(4):766-773. doi: 10.1097/GRF.0000000000000394. PMID 30204620
- [Background] Abo-Elroose AA, Ahmed MR, Shaaban MM, Ghoneim HM, Mohamed TY. Triple P with T-shaped lower segment suture; an effective novel alternative to hysterectomy in morbidly adherent anterior placenta previa. J Matern Fetal Neonatal Med. 2021 Oct;34(19):3187-3191. doi: 10.1080/14767058.2019.1678145. Epub 2019 Oct 15. PMID 31615304
- [Background] Di Mascio D, Cali G, D'antonio F. Updates on the management of placenta accreta spectrum. Minerva Ginecol. 2019 Apr;71(2):113-120. doi: 10.23736/S0026-4784.18.04333-2. Epub 2018 Nov 27. PMID 30486635